CLINICAL TRIAL: NCT07206654
Title: A Case-Control Study on the Presence, Causes, and Frequencies of Shoulder Girdle Musculoskeletal Complaints in Geriatrics With Diminished Vision
Brief Title: Prevalence and Determinants of Shoulder Girdle Musculoskeletal Complaints in Geriatric Patients With Diminished Vision
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Collaborators: Helwan University (Other)
Responsible Party: Principal Investigator, Mohamed Yasser Sayed Saif, Prof of Ophthalmology, Beni-Suef University
Other Study IDs: FMBSUREC/11022024/El Fayoumi
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Visual Impairment; Age-Related Macular Degeneration (AMD); Musculoskeletal Pain; Shoulder Pain; Geriatric Syndrome
Keywords: Geriatrics; Visual Impairment; Musculoskeletal Complaints; Shoulder Girdle
MeSH Terms: conditions — Vision Disorders; Macular Degeneration; Musculoskeletal Pain; Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group/Cohort 1: Cases (Elderly with visual impairment <6/60 due to AMD): Cases (Elderly with visual impairment <6/60 due to AMD)
- Group/Cohort 2: Controls (Elderly with normal vision, AMD-free): Controls (Elderly with normal vision, AMD-free)

SUMMARY:
This case-control study aims to investigate the prevalence and determinants of shoulder girdle musculoskeletal complaints (pain, spasm, stiffness, range of motion impairments) in geriatric patients (aged 60+) with diminished vision (visual acuity <6/60) due to Age-related Macular Degeneration (AMD), compared to a control group of age-matched elderly individuals with normal vision. The study will also assess the impact of these complaints on functional ability (Activities of Daily Living - ADL, Instrumental Activities of Daily Living - IADL) and quality of life using standardized questionnaires.

DETAILED DESCRIPTION:
This is an observational, case-control study conducted at the ophthalmology and geriatrics departments of Helwan University Hospitals and Beni-Suef University Hospitals. A total of 100 participants will be enrolled: 50 cases with visually significant AMD and visual acuity <6/60, and 50 controls with normal vision. All participants will undergo a comprehensive assessment including: detailed history taking, full ophthalmic examination (visual acuity, slit-lamp, fundus examination), geriatric assessment (ADL, IADL), and a structured musculoskeletal evaluation of the shoulder girdle and neck. The musculoskeletal evaluation will include assessment of pain (Visual Analog Scale), spasm, stiffness, and active/passive range of motion measured by an orthopedic surgeon using standardized tools like a digital inclinometer. Health-related quality of life will be measured using the Arabic Version of the National Eye Institute Visual Function Questionnaire (ARB-VFQ-25). Statistical analysis will be performed to compare the two groups and identify correlating factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 years or older.

For Case Group: Documented diagnosis of Age-Related Macular Degeneration (AMD) with visual impairment (visual acuity < 6/60).

For Control Group: Normal vision, free from AMD as diagnosed by fundus examination and Snellen test.

Exclusion Criteria:

* Musculoskeletal complaints due to Parkinsonism.

Musculoskeletal complaints due to Osteoarthritis (OA) or Multiple Sclerosis (MS).

Inability to provide informed consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study enrolled a total of 100 Egyptian geriatric participants, recruited from the ophthalmology and geriatrics clinics of Helwan University Hospitals and Beni-Suef University Hospitals.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-09-22 (Actual)

PRIMARY OUTCOMES:
Prevalence of Shoulder Girdle Pain | Singleassessmentatenrollment(Day1)
  Measure: Proportion of participants reporting shoulder girdle pain (Yes/No), assessed via standardized history and Visual Analog Scale (VAS).
Prevalence of Shoulder Girdle Spasm and Stiffness | Singleassessmentatenrollment(Day1)
  Measure: Proportion of participants with clinically identified shoulder girdle spasm and stiffness (Yes/No).

SECONDARY OUTCOMES:
Shoulder and Neck Range of Motion (ROM) | Singleassessmentatenrollment(Day1)
  Measure: Degrees of active and passive ROM (Flexion, Abduction, Internal/External Rotation) measured with a digital inclinometer. Impairment is defined as a positive difference between unaffected and affected shoulder.
Functional Status (ADL and IADL) | Singleassessmentatenrollment(Day1)
  Scores on the Groningen Activity Restriction Scale (GARS) for ADL and a standardized IADL questionnaire. Higher scores indicate more restrictions.
Vision-Related Quality of Life | Singleassessmentatenrollment(Day1)
  Composite score from the Arabic Version of the National Eye Institute Visual Function Questionnaire (ARB-VFQ-25). Higher scores indicate better quality of life
Reading Performance | Singleassessmentatenrollment(Day1)
  Reading distance (in cm) and required magnification power (X) for near tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Beni Suef University, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No